CLINICAL TRIAL: NCT07003945
Title: Clinical Outcomes of Percutaneous Intramyocardial Septal Radiofrequency Ablation Treating for Hypertrophic Obstructive Cardiomyopathy: A Large-Sample Study
Brief Title: Clinical Outcomes of PIMSRA Treating for Hypertrophic Obstructive Cardiomyopathy: A Large-Sample Study
Status: Active, not recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20242272-C-1
Record Dates: First submitted 2025-04-30; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-04

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy (HOCM)
Keywords: Cardiomyopathy, hypertrophic; Treatment outcome; safety; efficacy; Percutaneous intramyocardial septal radiofrequency ablation
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypertrophic Obstructive Cardiomyopathy Patients Underwent PIMSRA
  Interventions: Procedure: Percutaneous Intramyocardial Septal Radiofrequency Ablation

INTERVENTIONS:
Procedure: Percutaneous Intramyocardial Septal Radiofrequency Ablation — With the real-time guidance of TTE, a radiofrequency electrode needle was percutaneously inserted via the transapical intramyocardial approach into the hypertrophied septum for thermal ablation. Intraoperative TTE and 12-lead electrocardiographic monitoring were employed to assess the ablation extent and prevent vascular and cardiac conduction bundle injury. The success of ablation was confirmed by evaluating contrast medium perfusion defects in the ablated areas and comparing them with the preprocedural hypertrophied septum.

SUMMARY:
The Hypertrophic Cardiomyopathy Center of Xijing Hospital pioneered percutaneous intramyocardial septal radiofrequency ablation (PIMSRA) as an innovative treatment for hypertrophic obstructive cardiomyopathy (HOCM) to relieve left ventricular outflow tract obstruction. Clinical studies have confirmed PIMSRA's efficacy, safety and reliability, establishing it as a novel alternative for septal reduction therapy. As a novel interventional approach, comprehensive evaluation of its safety and therapeutic effectiveness is warranted.

Therefore, this retrospective study aims to:

* Investigate postoperative clinical outcomes and their influencing factors in HOCM patients undergoing PIMSRA;
* Analyze morphological and hemodynamic changes including: septal thickness, left ventricular outflow tract gradient, mid-ventricular pressure gradient and left ventricular flow field dynamics;
* Examine correlations between clinical/procedural parameters and clinical symptoms, quality of life and cardiac reverse remodeling indicators.

This study will provide high-quality evidence to support the clinical application of this novel procedure.

ELIGIBILITY:
Inclusion Criteria:

* All HOCM patients who underwent PIMSRA treatment, including those with left ventricular outflow tract and middle ventricular obstruction;
* Age from 18 to 90 years old.

Exclusion Criteria:

* Patients lost to follow-up whose follow-up period did not reach 6 months;
* Incomplete clinical data affected statistical analysis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with HOCM and with drug-refractory symptoms underwent PIMSRA in Xijing Hospital from 2016 to 2025.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | Observations were conducted from the immediate postoperative period through 1-year follow-up, with assessment time points including but not limited to 1 month, 3 months, 6 months, and 1 year.
  Major adverse cardiovascular events including but not limited to:
  1. All-cause death;
  2. Arrhythmic events: resuscitated cardiac arrest or ventricular tachycardia/fibrillation, appropriate implantable cardioverter-defibrillator discharge, atrioventricular block, pacemaker implantation and atrial fibrillation;
  3. Acute heart failure: acute pulmonary edema, new-onset NYHA class Ⅲ-IV symptoms, and heart failure-related hospitalization;
  4. Cardiogenic shock: cardiac disorder that results in a systolic blood pressure <90 mmHg for ≥30 min (or the need for vasopressors, inotropes or mechanical circulatory support to maintain systolic blood pressure ≥90 mmHg) with evidence of hypoperfusion;
  5. Severe systolic anterior motion: the proximal portion of the anterior mitral leaflet moved excessively close to the septum, resulting in extreme LVOT obstruction and acute haemodynamic collapse;
  6. Cerebrovascular events: all stroke (ischemic or hemorrhagic) and transient ischemic attacks.
Procedure-related adverse events | Observations were conducted from the immediate postoperative period through 1-year follow-up, with assessment time points including but not limited to 1 month, 3 months, 6 months, and 1 year.
  Any instrument or procedure-related complications, including but not limited to death, emergency surgery, pericardial tamponade requiring pericardiocentesis or surgery, bleeding, procedure-related stroke.
Interventricular septal thickness | Observations were conducted from the immediate postoperative period through 1-year follow-up, with assessment time points including but not limited to 1 month, 3 months, 6 months, and 1 year.
  Maximum septal thickness as measured by echocardiography.
Left ventricular outflow tract gradient | Observations were conducted from the immediate postoperative period through 1-year follow-up, with assessment time points including but not limited to 1 month, 3 months, 6 months, and 1 year.
  Left ventricular outflow tract gradient as measured by echocardiography.

SECONDARY OUTCOMES:
New York Heart Association Classification | Observations were conducted from the immediate postoperative period through 1-year follow-up, with assessment time points including but not limited to 1 month, 3 months, 6 months, and 1 year.
  The New York Heart Association Classification involved 4 classes. I-No limitation of physical activity, II-Slight limitation of physical activity, III-Marked limitation of physical activity, IV-Unable to carry on any physical activity without discomfort. A higher grade means worse heart function.
Kansas City Cardiomyopathy Questionnaire score | Observations were conducted from the immediate postoperative period through 1-year follow-up, with assessment time points including but not limited to 1 month, 3 months, 6 months, and 1 year.
  The Kansas City Cardiomyopathy Questionnaire was a 23-item, self-administered questionnaire that measure the participant's perception of their health status. It quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), quality of life (3 items) and social limitations (4 items). Scores were generated from each domain and scaled from 0 to 100, where lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life.
Late gadolinium enhancement | Observations were conducted from the immediate postoperative period through 1-year follow-up, with assessment time points including but not limited to 1 month, 3 months, 6 months, and 1 year.
  Late gadolinium enhancement measured by cardiac magnetic resonance.
Mean blood pressure | Observations were conducted from the immediate postoperative period through 1-year follow-up, with assessment time points including but not limited to 1 month, 3 months, 6 months, and 1 year.
  Mean systolic/diastolic blood pressure measured by ambulatory blood pressure monitoring.
Energy loss | Observations were conducted from the immediate postoperative period through 1-year follow-up, with assessment time points including but not limited to 1 month, 3 months, 6 months, and 1 year.
  Energy loss measured by vector flow mapping.

CONTACTS AND LOCATIONS:
Locations (1):
- Ultrasound Medicine Department of Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No